CLINICAL TRIAL: NCT01340209
Title: A Phase III Randomised, Double-blind, Placebo-controlled, Parallel-group Trial to Evaluate Safety and Efficacy of Tiotropium Inhalation Solution Delivered Via Respimat Inhaler (2.5 and 5 µg Once Daily) Compared With Placebo Over 52 Weeks in Patients With Moderate to Severe Persistent Asthma
Brief Title: Evaluation of Tiotropium 2.5 and 5 µg Once Daily Delivered Via the Respimat Inhaler Compared to Placebo in Patient With Moderate to Severe Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.464
Record Dates: First submitted 2011-04-13; First posted 2011-04-22 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — tiotropium-olodaterol

ARMS (3):
- Tiotropium Respimat (low dose) (Experimental): Tiotropium low dose once daily delivered with Respimat inhaler
  Interventions: Drug: Tiotropium Respimat
- Tiotropium Respimat (high dose) (Experimental): Tiotropium high dose once daily delivered with Respimat inhaler
  Interventions: Drug: Tiotropium Respimat
- Placebo Respimat (Placebo Comparator): Tiotropium placebo once daily delivered with Respimat inhaler
  Interventions: Drug: Placebo Respimat

INTERVENTIONS:
Drug: Tiotropium Respimat — Tiotropium high dose once daily delivered with Respimat inhaler
  Arms: Tiotropium Respimat (high dose)
Drug: Placebo Respimat — Tiotropium placebo once daily delivered with Respimat inhaler
  Arms: Placebo Respimat
Drug: Tiotropium Respimat — Tiotropium low dose once daily delivered with Respimat inhaler
  Arms: Tiotropium Respimat (low dose)

SUMMARY:
The aim of this trial is to evaluate the safety and efficacy of 2.5 and 5 µg tiotropium over a 52-week treatment period as compared to placebo. Tiotropium inhalation solution delivered by the Respimat inhaler will be examined on top of maintenance treatment with inhaled corticosteroid controller medication in patients with moderate to severe persistent asthma. Efficacy and safety will be assessed by measuring effects on lung function, effects on asthma exacerbations, effects on asthma control, and number of adverse events.

ELIGIBILITY:
Inclusion criteria:

1. All patients including the patients under age (under 20 years old) must sign and date an Informed Consent Form consistent with ICH-GCP guidelines and Good Clinical Practice (GCP) prior to participation in the trial [i.e. prior to any trial procedures, including any pre-trial washout of medications and medication restrictions for pulmonary function test (PFT) at Visit 1]. Regarding patients under age, a guardian or a legally authorised representative must also sign and date an Informed Consent Form.
2. Male or female outpatients aged at least 18 years but not more than 75 years at Visit 0.
3. All patients must have at least a 12-week history of asthma at the time of enrolment (Visit 0) into the trial. The diagnosis should be confirmed at Visit 1 by fulfilling inclusion criterion 5.
4. The initial diagnosis of asthma must have been made before the patient's age of 40.
5. The diagnosis of asthma has to be confirmed at Visit 1 with a bronchodilator reversibility (15-30 minutes after 400 µg salbutamol) resulting in a Forced Expiratory Volume in one second (FEV1) increase of at least 12% and at least 200 mL .
6. All patients must have been on maintenance treatment with a medium, stable dose of inhaled corticosteroids (ICS) [alone or in a fixed combination with a Long-acting beta-adrenergic (LABA)] for at least 4 weeks prior to Visit 1.
7. All patients must be symptomatic at Visit 1 (screening) and prior to randomisation at Visit 2 as defined by an Asthma Control Questionnaire (ACQ) mean score of at least 1.5.
8. All patients must have a pre-bronchodilator FEV1 at least 60% and less than or equal to 90% of predicted normal at Visit 1.
9. Patients must be never-smokers or ex-smokers who stopped smoking at least one year (52 weeks) prior to enrolment (Visit 0) and who have a smoking history of less than 10 pack years.
10. Patients must be able to use the Respimat inhaler correctly, which is judged at the discretion of the investigator..
11. Patients must be able to perform all trial related procedures including technically acceptable PFTs and use of electronic diary (eDiary)/peak flow meter, which is judged at the discretion of the investigator.

Exclusion criteria:

1. Patients with a significant disease other than asthma. A significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the trial, or (ii) influence the results of the trial, or (iii) cause concern regarding the patient's ability to participate in the trial.
2. Patients with a clinically relevant abnormal screening (Visit 1) haematology or blood chemistry if the abnormality defines a significant disease as defined in exclusion criterion no 1.
3. Patients with a recent history (i.e. 6 months or less) of myocardial infarction prior to Visit 0.
4. Patients who have been hospitalised for cardiac failure during the past year prior to Visit 0.
5. Patients with any unstable or life-threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year prior to Visit 0.
6. Patients with lung diseases other than asthma (e.g. COPD).
7. Patients with known active tuberculosis.
8. Patients with malignancy and/or patients who have undergone resection, radiation therapy or chemotherapy for malignancy within the last 5 years prior to Visit 0. Patients with treated basal cell carcinoma are allowed.
9. Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criterion no. 1.
10. Patients with significant alcohol or drug abuse, which is judged at the discretion of the investigator, within the past 2 years prior to Visit 0.
11. Patients with known hypersensitivity to anticholinergic drugs, benzalkonium chloride (BAC), ethylenediaminetetraacetic acid (EDTA), or any other components of the study medication delivery systems.
12. Pregnant or nursing women.
13. Women of childbearing potential not using a highly effective method of birth control.
14. Patients who have taken an investigational drug within 4 weeks prior to Visit 1.
15. Patients who have been treated with beta-blocker medication within four weeks prior to Visit 1 and/or during the screening period. Topical cardio-selective beta-blocker eye medications for non-narrow angle glaucoma are allowed.
16. Patients who have been treated with the long-acting anticholinergic tiotropium (Spiriva) within four weeks prior to Visit 1 and/or during the screening period.
17. Patients who have been treated with oral beta-adrenergics within four weeks prior to Visit 1 and/or during the Screening period.
18. Patients who have been treated with systemic corticosteroids within four weeks prior to Visit 1 and/or during the screening period.
19. Patients who have been treated with anti-IgE antibodies, e.g. omalizumab (Xolair®), within 6 months prior to Visit 1 and/or during the screening period.
20. Patients who have been treated with other non-approved and according to international guidelines not recommended "experimental" drugs for routine asthma therapy within four weeks prior to Visit 1 and/or during the screening period.
21. Patients with any asthma exacerbation or any respiratory tract infection in the four weeks prior to Visit 1 and/or during the screening period.
22. Patients who are currently participating in another trial.
23. Patients with narrow-angle glaucoma and/or micturition disorder due to prostatic hyperplasia.
24. Patients with below 80% of the eDiary completion compliance on Visit 2 (diary compliance of at least 80% is required).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (55):
- Japan (55):
  - 205.464.81020 Boehringer Ingelheim Investigational Site, Asahikawa, Hokkaido
  - 205.464.81031 Boehringer Ingelheim Investigational Site, Atsugi, Kanagawa
  - 205.464.81029 Boehringer Ingelheim Investigational Site, Chigasaki, Kanagawa
  - 205.464.81011 Boehringer Ingelheim Investigational Site, Chino, Nagano
  - 205.464.81050 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 205.464.81051 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 205.464.81006 Boehringer Ingelheim Investigational Site, Edogawa-ku, Tokyo
  - 205.464.81010 Boehringer Ingelheim Investigational Site, Fujisawa, Kanagawa
  - 205.464.81016 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 205.464.81004 Boehringer Ingelheim Investigational Site, Hanno, Saitama
  - 205.464.81040 Boehringer Ingelheim Investigational Site, Himeji, Hyogo
  - 205.464.81041 Boehringer Ingelheim Investigational Site, Himeji, Hyogo
  - 205.464.81053 Boehringer Ingelheim Investigational Site, Himeji, Hyogo
  - 205.464.81007 Boehringer Ingelheim Investigational Site, Hino, Tokyo
  - 205.464.81015 Boehringer Ingelheim Investigational Site, Hiroshima, Hiroshima
  - 205.464.81002 Boehringer Ingelheim Investigational Site, Hitachinaka, Ibaraki
  - 205.464.81048 Boehringer Ingelheim Investigational Site, Iizuka, Fukuoka
  - 205.464.81005 Boehringer Ingelheim Investigational Site, Itabashi-ku, Tokyo
  - 205.464.81033 Boehringer Ingelheim Investigational Site, Kaga, Ishikawa
  - 205.464.81017 Boehringer Ingelheim Investigational Site, Kagoshima, Kagoshima
  - 205.464.81023 Boehringer Ingelheim Investigational Site, Kamogawa, Chiba
  - 205.464.81024 Boehringer Ingelheim Investigational Site, Kisarazu, Chiba
  - 205.464.81047 Boehringer Ingelheim Investigational Site, Kitakyusyu,Fukuoka
  - 205.464.81008 Boehringer Ingelheim Investigational Site, Kiyose, Tokyo
  - 205.464.81046 Boehringer Ingelheim Investigational Site, Kochi, Kochi
  - 205.464.81025 Boehringer Ingelheim Investigational Site, Kodaira, Tokyo
  - 205.464.81022 Boehringer Ingelheim Investigational Site, Koshigaya, Saitama
  - 205.464.81043 Boehringer Ingelheim Investigational Site, Kurashiki, Okayama
  - 205.464.81044 Boehringer Ingelheim Investigational Site, Kure, Hiroshima
  - 205.464.81014 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 205.464.81038 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 205.464.81003 Boehringer Ingelheim Investigational Site, Maebashi, Gumma
  - 205.464.81042 Boehringer Ingelheim Investigational Site, Matsue, Shimane
  - 205.464.81026 Boehringer Ingelheim Investigational Site, Minato-ku, Tokyo
  - 205.464.81012 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 205.464.81013 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 205.464.81034 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 205.464.81035 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 205.464.81036 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 205.464.81037 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 205.464.81001 Boehringer Ingelheim Investigational Site, Obihiro, Hokkaido
  - 205.464.81018 Boehringer Ingelheim Investigational Site, Obihiro, Hokkaido
  - 205.464.81054 Boehringer Ingelheim Investigational Site, Oita, Oita
  - 205.464.81055 Boehringer Ingelheim Investigational Site, Oita, Oita
  - 205.464.81039 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 205.464.81049 Boehringer Ingelheim Investigational Site, Saga, Saga
  - 205.464.81019 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 205.464.81021 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 205.464.81027 Boehringer Ingelheim Investigational Site, Setagaya-Ku, Tokyo
  - 205.464.81028 Boehringer Ingelheim Investigational Site, Setagaya-ku, Tokyo
  - 205.464.81045 Boehringer Ingelheim Investigational Site, Toon, Ehime
  - 205.464.81009 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa
  - 205.464.81052 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa
  - 205.464.81030 Boehringer Ingelheim Investigational Site, Yokosuka, Kanagawa
  - 205.464.81032 Boehringer Ingelheim Investigational Site, Zama

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Halpin DMG, Meltzer EO, Pisternick-Ruf W, Moroni-Zentgraf P, Engel M, Zaremba-Pechmann L, Casale T, FitzGerald JM. Peak expiratory flow as an endpoint for clinical trials in asthma: a comparison with FEV1. Respir Res. 2019 Jul 18;20(1):159. doi: 10.1186/s12931-019-1119-6. PMID 31319851
- [Derived] Ohta K, Ichinose M, Tohda Y, Engel M, Moroni-Zentgraf P, Kunimitsu S, Sakamoto W, Adachi M. Long-Term Once-Daily Tiotropium Respimat(R) Is Well Tolerated and Maintains Efficacy over 52 Weeks in Patients with Symptomatic Asthma in Japan: A Randomised, Placebo-Controlled Study. PLoS One. 2015 Apr 20;10(4):e0124109. doi: 10.1371/journal.pone.0124109. eCollection 2015. PMID 25894430

RESULTS

PARTICIPANT FLOW:
Groups:
- Tiotropium Respimat (2.5 µg): Tiotropium Respimat: Tiotropium 2.5 µg once daily delivered with Respimat inhaler
- Tiotropium Respimat (5 μg): Tiotropium Respimat: Tiotropium 5 μg once daily delivered with Respimat inhaler
Period: Overall Study
Arm/Group | Placebo Respimat | Tiotropium Respimat (2.5 µg) | Tiotropium Respimat (5 μg)
Started | 57 | 114 | 114
Completed | 52 | 106 | 106
Not Completed | 5 | 8 | 8
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Protocol Violation | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Other reason not defined above | 3 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Respimat | Tiotropium Respimat (2.5 µg) | Tiotropium Respimat (5 μg) | Total
Number analyzed (Participants) | 57 | 114 | 114 | 285
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (13.0) | 44.7 (12.1) | 42.6 (12.8) | 44.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 72 | 66 | 176
  Male | 19 | 42 | 48 | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Drug-related Adverse Events
Description: The primary endpoint is the number of patients with drug-related adverse events
Time Frame: after the first dose of trial medication and within 30 days after the last dose of trial medication, up to 409
Population: Treated set: all randomised patients who received at least 1 dose of study medication
Measure: Number; unit: participants
Arm/Group | Placebo Respimat | Tiotropium Respimat (2.5 µg) | Tiotropium Respimat (5 μg)
Number analyzed (Participants) | 57 | 114 | 114
participants | 3 | 6 | 10

2. Secondary Outcome: Trough FEV1 Response
Description: Trough FEV1 response was defined as change from baseline at week 52
Time Frame: baseline and week 52
Population: Full analysis set: all patients of the treated set for which baseline and at least 1 post-baseline efficacy measurement were available
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo Respimat | Tiotropium Respimat (2.5 µg) | Tiotropium Respimat (5 μg)
Number analyzed (Participants) | 56 | 114 | 114
Liter | 0.075 (0.039) | 0.087 (0.027) | 0.187 (0.027)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tiotropium Respimat (2.5 µg); Difference calculated as Tiotropium 2.5 µg minus placebo; Test type: Superiority or Other; p = 0.7971, Mixed Models Analysis; adjusted for treatment, week, baseline, treatment*week and baseline*week; Mean Difference (Final Values) = 0.012, 95% CI 2-sided [-0.082 to 0.106], Standard Error of Mean 0.048
Statistical Analysis 2: Comparison: Placebo Respimat vs Tiotropium Respimat (5 μg); Difference calculated as Tiotropium 5 μg minus placebo; Test type: Superiority or Other; p = 0.0203, Mixed Models Analysis; adjusted for treatment, week, baseline, treatment*week and baseline*week; Mean Difference (Final Values) = 0.112, 95% CI 2-sided [0.018 to 0.207], Standard Error of Mean 0.048

3. Secondary Outcome: Trough FVC Response
Description: Trough FVC response was defined as change from baseline at week 52
Time Frame: baseline and week 52
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo Respimat | Tiotropium Respimat (2.5 µg) | Tiotropium Respimat (5 μg)
Number analyzed (Participants) | 56 | 114 | 114
Liter | 0.122 (0.044) | 0.085 (0.030) | 0.204 (0.031)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tiotropium Respimat (2.5 µg); Difference calculated as Tiotropium 2.5 µg minus placebo; Test type: Superiority or Other; p = 0.4944, Mixed Models Analysis; adjusted for treatment, week, baseline, treatment*week and baseline*week; Mean Difference (Final Values) = -0.037, 95% CI 2-sided [-0.141 to 0.068], Standard Error of Mean 0.053
Statistical Analysis 2: Comparison: Placebo Respimat vs Tiotropium Respimat (5 μg); Difference calculated as Tiotropium 5 μg minus placebo; Test type: Superiority or Other; p = 0.1270, Mixed Models Analysis; adjusted for treatment, week, baseline, treatment*week and baseline*week; Mean Difference (Final Values) = 0.082, 95% CI 2-sided [-0.023 to 0.188], Standard Error of Mean 0.054

4. Secondary Outcome: Trough PEF Response
Description: Trough PEF response was defined as change from baseline at week 52
Time Frame: baseline and week 52
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo Respimat | Tiotropium Respimat (2.5 µg) | Tiotropium Respimat (5 μg)
Number analyzed (Participants) | 56 | 114 | 114
L/min | 35.078 (10.119) | 35.576 (6.917) | 69.254 (7.004)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tiotropium Respimat (2.5 µg); Difference calculated as Tiotropium 2.5 µg minus placebo; Test type: Superiority or Other; p = 0.9677, Mixed Models Analysis; adjusted for treatment, week, baseline, treatment*week and baseline*week; Mean Difference (Final Values) = 0.498, 95% CI 2-sided [-23.634 to 24.630], Standard Error of Mean 12.282
Statistical Analysis 2: Comparison: Placebo Respimat vs Tiotropium Respimat (5 μg); Difference calculated as Tiotropium Respimat 5 μg minus placebo; Test type: Superiority or Other; p = 0.0058, Mixed Models Analysis; adjusted for treatment, week, baseline, treatment*week and baseline*week; Median Difference (Final Values) = 34.176, 95% CI 2-sided [9.919 to 58.432], Standard Error of Mean 12.346

5. Secondary Outcome: Weekly Mean PEFam Response
Description: Weekly mean PEFam response was defined as change from baseline at week 52
Time Frame: baseline and week 52
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo Respimat | Tiotropium Respimat (2.5 µg) | Tiotropium Respimat (5 μg)
Number analyzed (Participants) | 56 | 114 | 114
L/min | 2.288 (7.554) | 10.934 (5.231) | 8.504 (5.267)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tiotropium Respimat (2.5 µg); Difference calculated as Tiotropium 2.5 µg minus placebo; Test type: Superiority or Other; p = 0.3468, Mixed Models Analysis; adjusted for treatment, week, baseline, treatment*week and baseline*week; Mean Difference (Final Values) = 8.646, 95% CI 2-sided [-9.388 to 26.680], Standard Error of Mean 9.182
Statistical Analysis 2: Comparison: Placebo Respimat vs Tiotropium Respimat (5 μg); Difference calculated as Tiotropium 5 μg minus placebo; Test type: Superiority or Other; p = 0.5013, Mixed Models Analysis; adjusted for treatment, week, baseline, treatment*week and baseline*week; Mean Difference (Final Values) = 6.216, 95% CI [-11.927 to 24.359], Standard Error of Mean 9.238

6. Secondary Outcome: Weekly Mean PEFpm Response
Description: Weekly mean PEFpm response was defined as change from baseline at week 52
Time Frame: baseline and week 52
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo Respimat | Tiotropium Respimat (2.5 µg) | Tiotropium Respimat (5 μg)
Number analyzed (Participants) | 56 | 114 | 114
L/min | -10.357 (7.566) | 1.101 (5.239) | 6.041 (5.284)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tiotropium Respimat (2.5 µg); Difference calculated as Tiotropium 2.5 µg minus placebo; Test type: Superiority or Other; p = 0.2132, Mixed Models Analysis; adjusted for treatment, week, baseline, treatment*week and baseline*week; Mean Difference (Final Values) = 11.458, 95% CI 2-sided [-6.601 to 29.517], Standard Error of Mean 9.196
Statistical Analysis 2: Comparison: Placebo Respimat vs Tiotropium Respimat (5 μg); Difference calculated as Tiotropium 5 μg minus placebo; Test type: Superiority or Other; p = 0.0766, Mixed Models Analysis; adjusted for treatment, week, baseline, treatment*week and baseline*week; Mean Difference (Final Values) = 16.398, 95% CI 2-sided [-1.759 to 34.555], Standard Error of Mean 9.245

7. Secondary Outcome: Weekly Mean PEF Variability Response
Description: Weekly mean PEF variability response was defined as change from baseline at week 52.
  The PEF variability is the absolute difference between morning and evening PEF value, divided by their mean, expressed as a percent. Response was defined as change from baseline.
Time Frame: baseline and week 52
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Placebo Respimat | Tiotropium Respimat (2.5 µg) | Tiotropium Respimat (5 μg)
Number analyzed (Participants) | 56 | 114 | 114
percentage | -0.367 (0.851) | -0.968 (0.595) | 0.197 (0.595)
Statistical Analysis 1: Comparison: Placebo Respimat vs Tiotropium Respimat (2.5 µg); Difference calculated as Tiotropium 2.5 µg minus placebo; Test type: Superiority or Other; p = 0.5629, Mixed Models Analysis; adjusted for treatment, week, baseline, treatment*week and baseline*week; Mean Difference (Final Values) = -0.601, 95% CI 2-sided [-2.637 to 1.436], Standard Error of Mean 1.038
Statistical Analysis 2: Comparison: Placebo Respimat vs Tiotropium Respimat (5 μg); Difference calculated as Tiotropium 5 μg minus placebo; Test type: Superiority or Other; p = 0.5871, Mixed Models Analysis; adjusted for treatment, week, baseline, treatment*week and baseline*week; Mean Difference (Final Values) = 0.564, 95% CI 2-sided [-1.473 to 2.601], Standard Error of Mean 1.038

8. Secondary Outcome: Weekly Mean Number of Puffs of Rescue Medication During the Whole Day (Response)
Description: Response of weekly mean number of puffs of rescue medication during the whole day at week 52. Response was defined as change from baseline.
Time Frame: baseline and week 52
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Puffs
Arm/Group | Placebo Respimat | Tiotropium Respimat (2.5 µg) | Tiotropium Respimat (5 μg)
Number analyzed (Participants) | 50 | 105 | 103
Puffs | -0.25 (0.77) | -0.29 (1.01) | -0.22 (0.96)

9. Secondary Outcome: Weekly Mean Score of Asthma Symptoms in the Morning (Response)
Description: Response of weekly mean score of asthma symptoms in the morning at week 52. Response was defined as change from baseline.
  5-point verbal rating scale, with answer 1 representing no impairment at all and answer 5 representing the greatest impairment.
Time Frame: baseline and week 52
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Respimat | Tiotropium Respimat (2.5 µg) | Tiotropium Respimat (5 μg)
Number analyzed (Participants) | 50 | 103 | 103
Scores on a scale | -0.22 (0.43) | -0.14 (0.49) | -0.21 (0.43)

10. Secondary Outcome: Weekly Mean Score of Asthma Symptoms During the Day (Response)
Description: Response of weekly mean score of asthma symptoms during the day at week 52. Response was defined as change from baseline.
  5-point verbal rating scale, with answer 1 representing no impairment at all and answer 5 representing the greatest impairment.
Time Frame: baseline and week 52
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo Respimat | Tiotropium Respimat (2.5 µg) | Tiotropium Respimat (5 μg)
Number analyzed (Participants) | 50 | 105 | 103
Scores on a scale | -0.24 (0.35) | -0.15 (0.48) | -0.17 (0.48)

ADVERSE EVENTS:
Time Frame: after the first dose of trial medication and within 30 days after the last dose of trial medication, up to 409 days
Arm/Group | Placebo Respimat | Tiotropium Respimat (2.5 µg) | Tiotropium Respimat (5 μg)
Serious Adverse Events (participants affected / at risk) | 9/57 | 4/114 | 4/114
Other Adverse Events (participants affected / at risk) | 50/57 | 97/114 | 101/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Respimat (N=57) | Tiotropium Respimat (2.5 µg) (N=114) | Tiotropium Respimat (5 μg) (N=114)
Mesenteric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1
Cyst (General disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Respimat (N=57) | Tiotropium Respimat (2.5 µg) (N=114) | Tiotropium Respimat (5 μg) (N=114)
Constipation (Gastrointestinal disorders) | 3 | 0 | 1
Gastritis (Gastrointestinal disorders) | 4 | 3 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 6
Bronchitis (Infections and infestations) | 4 | 15 | 11
Gastroenteritis (Infections and infestations) | 3 | 4 | 12
Influenza (Infections and infestations) | 2 | 6 | 5
Nasopharyngitis (Infections and infestations) | 24 | 51 | 55
Pharyngitis (Infections and infestations) | 2 | 15 | 9
Upper respiratory tract infection (Infections and infestations) | 2 | 8 | 5
Ligament sprain (Injury, poisoning and procedural complications) | 3 | 2 | 3
Peak expiratory flow rate decreased (Investigations) | 12 | 9 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 4
Headache (Nervous system disorders) | 1 | 7 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 21 | 34 | 32
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 7
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.